CLINICAL TRIAL: NCT00557206
Title: Multicenter Phase II Trial of Oxaliplatin and Docetaxel for Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck
Brief Title: Oxaliplatin and Docetaxel for Recurrent or Metastatic Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was terminated
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Balkrishna Jahagirdar, Principal Investigator, Minneapolis Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX-04-033; VA-CORNET
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Neoplasms; Head and Neck Neoplasms
Keywords: Recurrent Disease; Metastatic Disease; Squamous Cell Carcinoma; Multicenter; Phase II
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms; Recurrence; Neoplasm Metastasis; Carcinoma, Squamous Cell | interventions — Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This is a single arm trial.
  Interventions: Drug: Oxaliplatin and Docetaxel

INTERVENTIONS:
Drug: Oxaliplatin and Docetaxel — Chemotherapy
  Oxaliplatin 130mg/m2 on day 1; and Docetaxel 75mg/m2 on day 1; every 21 days.

SUMMARY:
Patient receiving oxaliplatin and docetaxel will have longer progression free survival than those patients receiving standard care.

DETAILED DESCRIPTION:
Oxaliplatin: 130mg/m2 given on day 1 by intravenous injection; and Docetaxel: 60mg/m2 given on day 1 by intravenous injection

Cycles are repeated every 21 days until disease progression, unacceptable toxicity or subject's withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or locoregionally recurrent SCCHN deemed incurable by local therapy
* Measureable disease
* No prior use of palliative chemo after the SCCHN is deemed incurable by local therapy
* No prior treatment with oxaliplatin or docetaxel
* 18 years of age or older
* ECOG Performance status 0-1
* ANC 1,500/mcl or greater
* Adequate renal function
* Adequate liver function
* Recovered from acute and late effects of any prior treatment with a minimum of 4 weeks from the last session to enrollment in the study
* Patient or their legal representative must be able to read, understand, and provide informed consent
* Patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication

Exclusion Criteria:

* Patients with an active documented infection or with a fever (38.5 degrees celsius or higher) within 3 days of the first scheduled dose of study treatment
* Patients with active CNS metastases
* Hypercalcemia related to SCCHN
* History of prior malignancy with the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intraepithelial neoplasia or localized prostate cancer
* Patients with known hypersensitivity to any of the components of oxaliplatin or docetaxel or to other drugs formulated with polysorbate 90
* Patients receiving concurrent investigational therapy or investigational therapy less than 30 days from first scheduled dose of study therapy
* Peripheral neuropathy grade 2 or higher
* Any medical condition deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
* History of allogeneic transplant
* Known HIV or Hepatitis B or C (active, previously treated or both)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Response rate as determined by RECIST criteria every 6 weeks. | 2 Years

SECONDARY OUTCOMES:
Toxicity and Quality of Life assessments every 3 weeks. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Balkrishna Jahagirdar, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center; Vicki A Morrison, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- VA Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Degardin M, Cappelaere P, Krakowski I, Fargeot P, Cupissol D, Brienza S. Phase II trial of oxaliplatin (L-OHP) in advanced, recurrent and/or metastatic squamous cell carcinoma of the head and neck. Eur J Cancer B Oral Oncol. 1996 Jul;32B(4):278-9. doi: 10.1016/0964-1955(95)00082-8. No abstract available. PMID 8776427
- [Background] Ibrahim A, Hirschfeld S, Cohen MH, Griebel DJ, Williams GA, Pazdur R. FDA drug approval summaries: oxaliplatin. Oncologist. 2004;9(1):8-12. doi: 10.1634/theoncologist.9-1-8. PMID 14755010
- [Background] Grothey A. Oxaliplatin-safety profile: neurotoxicity. Semin Oncol. 2003 Aug;30(4 Suppl 15):5-13. doi: 10.1016/s0093-7754(03)00399-3. PMID 14523789
- [Background] Rixe O, Ortuzar W, Alvarez M, Parker R, Reed E, Paull K, Fojo T. Oxaliplatin, tetraplatin, cisplatin, and carboplatin: spectrum of activity in drug-resistant cell lines and in the cell lines of the National Cancer Institute's Anticancer Drug Screen panel. Biochem Pharmacol. 1996 Dec 24;52(12):1855-65. doi: 10.1016/s0006-2952(97)81490-6. PMID 8951344
- [Background] Kollmannsberger C, Rick O, Derigs HG, Schleucher N, Schoffski P, Beyer J, Schoch R, Sayer HG, Gerl A, Kuczyk M, Spott C, Kanz L, Bokemeyer C. Activity of oxaliplatin in patients with relapsed or cisplatin-refractory germ cell cancer: a study of the German Testicular Cancer Study Group. J Clin Oncol. 2002 Apr 15;20(8):2031-7. doi: 10.1200/JCO.2002.08.050. PMID 11956262
- [Background] Dieras V, Bougnoux P, Petit T, Chollet P, Beuzeboc P, Borel C, Husseini F, Goupil A, Kerbrat P, Misset JL, Bensmaine MA, Tabah-Fisch I, Pouillart P. Multicentre phase II study of oxaliplatin as a single-agent in cisplatin/carboplatin +/- taxane-pretreated ovarian cancer patients. Ann Oncol. 2002 Feb;13(2):258-66. doi: 10.1093/annonc/mdf018. PMID 11886003